CLINICAL TRIAL: NCT07228611
Title: Comparison of Osteoporosis Risk in the Subacute and Chronic Periods Following Stroke and Evaluation of Factors Increasing Osteoporosis
Brief Title: Assesment and Comparison of Osteoporosis Risk Factors After Stroke
Status: Recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Naz Kalem, PM&R Specialist, Ankara Etlik City Hospital
Other Study IDs: AEŞH-BADEK-2025-478
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Stroke Osteoporosis
MeSH Terms: interventions — Bone Density

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Subacute Stroke
  Interventions: Diagnostic Test: Bone Mineral Density
- Chronic Stroke
  Interventions: Diagnostic Test: Bone Mineral Density
- Healthy Volunteer
  Interventions: Diagnostic Test: Bone Mineral Density

INTERVENTIONS:
Diagnostic Test: Bone Mineral Density — Patients who have had a stroke and are at risk of fracture, and for whom routine assessment requires Bone Mineral Density (BMD) testing, will be included in the study. In addition, patients who have already undergone BMD testing for osteoporosis screening and who present to the outpatient clinic, with similar age and comorbidities, will be screened from the system, and 28 non-stroke patients who agree to participate will be included in the study.

SUMMARY:
The aim of this study is to evaluate the effect of these factors and stroke itself on osteoporosis developing after stroke. Thus, the expected benefit of the study is to contribute to the identification and determination of the need for treatment in high-risk patients through further studies. There are no expected risks from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Followed by ischemic or hemorrhagic stroke
2. Between 1 week and 6 months or >1 year has passed since the date of the event
3. Being between 55 and 85 years of age

Exclusion Criteria:

1. The patient has additional neurological conditions besides stroke
2. The patient has a psychiatric condition
3. History of recurrent stroke
4. BMD scan performed within the last year for stroke patients
5. Having received osteoporosis treatment before or after the stroke
6. The patient having a fragility fracture before the stroke
7. The patient having a hip fracture or hip prosthesis
8. The patient having an additional condition that affects physical function before the stroke (amputation, severe fracture)
9. The patient has an additional disease or medication use that could cause secondary osteoporosis
10. The patient's stroke did not cause physical function loss

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fifty-six stroke patients receiving inpatient treatment will be evaluated. In addition, patients who have visited the outpatient clinic and have already undergone BMD scanning for osteoporosis screening, with similar age and comorbidities, will be screened from the system, and 28 non-stroke patients who agree to participate will be randomly included in the study.
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Bone Mineral Density | First day of hospitalization

SECONDARY OUTCOMES:
Brunnstrom | First day of hospitalization
Modified Barthel Index | First day of hospitalization
Modified Ashworth Scale | First day of hospitalization
Modified Fall Impact Scale | First day of hospitalization
Vitamin D, prealbumin, and albumin | First day of hospitalization
Baseline Digital Hand Dynamometer 198 LB/90 kg | First day of hospitalization
  Patients' muscle strength will be measured using a Baseline Digital Hand Dynamometer at 198 LB/90 kg for both the dominant and non-dominant extremities.
Measurements of quadriceps muscle thickness and biceps muscle thickness | First day of hospitalization
  Regional sarcopenia of the plegic and non-plegic extremities will also be assessed using the STAR formula with measurements of anterior thigh muscle thickness and anterior arm muscle thickness by ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)